CLINICAL TRIAL: NCT00271882
Title: PTSD and Risk Behavior in HIV Positive Female Adolescents
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 053
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: PTSD; Sexual Abuse; HIV Infections
Keywords: Adolescent Females; HIV positive; PTSD; Sexual Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; HIV Infections; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a qualitative study using a purposive sampling methodology to interview HIV-positive female adolescents who have experienced physical and/or sexual abuse. An open-ended, in-depth interview, occurring over one to two sessions, will be conducted with each participant.

DETAILED DESCRIPTION:
This study is expected to take approximately 12 months to accrue participants and complete all the interviews. The interview will be conducted in one or two sessions and will be up to two hours in duration per session.

The study will initially be conducted at three ATN clinical sites with approximately 20 females recruited per site for a total of 60 participants. Other ATN clinical sites may be allowed to participate in the future if the study is slow to accrue.

The participants consist of English speaking women, ages 18-24 years, who acquired HIV through heterosexual intercourse or injection drug use after the age of 9 years, reported a history of sexual and/or physical abuse prior to age 18, and engaged in vaginal or anal intercourse in the 4 months prior to screening.

Approximately half of the participants will report a recent history of substance use as defined by study criteria and approximately half of the participants will report no such history.

Eligible patients will be identified and screened by the ATN research staff at the participating sites. The Protocol Chair and trained Research Assistant will conduct the open-ended qualitative interviews using an open-ended script. The interview will be audio-taped and transcribed. Prior to the open-ended script interview, participants will be asked about Posttraumatic Stress Disorder symptoms, abuse history, substance use, sexual behavior, and demographics. Responses to these questions will not be audio-taped and will be entered into the ATN 053 database by the ATN site staff.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 24 years old, inclusive, at the time of administration of the Screening Questionnaire.
* Female birth gender
* Verbal confirmation of acquisition of behaviorally-acquired HIV infection including from injection drug use (IDU) or heterosexual intercourse (vaginal, oral and/or anal) after the age of 9 years
* HIV-1 infection as documented by a positive result on any of the following licensed tests at any time: any antibody test confirmed by Western blot, HIV culture, plasma HIV-1 RNA PCR > 1,000 copies/mL or a HIV DNA PCR
* History of physical and/or sexual abuse prior to age 18 years old documented by a Screening Questionnaire
* Voluntary vaginal and/or anal intercourse with a male within the 4 months prior to screening.
* Ability to understand and communicate in spoken English sufficient to provide informed consent and to be interviewed
* Availability of enrollment slots for the participant's assigned substance-use category at the time of the Screening Questionnaire. (Approximately half of the participants will report substance use) This will be monitored throughout the study enrollment period.
* Willingness to have the qualitative study interview audio-taped
* Willingness and ability to provide informed consent

Exclusion Criteria:

* Currently suicidal or homicidal by clinician judgment
* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood, exhibiting manic, suicidal, or violent behavior);
* Visibly intoxicated or under the influence of psychoactive agents; or
* Presents as acutely ill.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: English speaking women, 18-24 years old with behaviorally- acquired HIV through heterosexual intercourse or injection drug use after the age of 9 years, who report a history of sexual and/or physical abuse prior to age 18, and who have engaged in vaginal or anal intercourse in the 4 months prior to screening.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Explore the interrelationship between abuse and sexual risk behavior | 12 Months
  To explore the interrelationship between abuse and sexual risk behavior in behaviorally-acquired HIV-positive female adolescents who report abuse histories
Explore the interrelationship between abuse, substance use and sexual risk behavior | 12 Months
  To explore the interrelationship between abuse, substance use and sexual risk behavior in those participants who meet substance use criteria

SECONDARY OUTCOMES:
Assess preferred intervention delivery strategies for an abuse-related intervention | 12 Months
  To assess preferred intervention delivery strategies for an abuse-related intervention such as length of treatment, incorporation of support/guardian figure, incorporation of issues related to HIV, and incorporation of specific sexual risk behavior modules.
Identify strengths/protective factors | 12 Months
  To identify strengths/protective factors (coping strategies, parent or network support) in girls who have experienced abuse that may be utilized to enhance the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Clum, Ph.D, Study Chair — Tulane School of Public Health and Tropical Medicine
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Montefiore Medical Center, The Bronx, New York
  - The Children's Hosp. of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org